CLINICAL TRIAL: NCT06843213
Title: Teaching Harm Reduction in Vulnerable Environments (THRIVE): A Peer-led Intervention Bridging Acute Care Settings and the Discharge to the Community
Brief Title: Teaching Harm Reduction in a Hospital Setting: A Peer-led Intervention
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 857581; 1R01DA057633 (NIH)
Record Dates: First submitted 2025-01-13; First posted 2025-02-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder; Harm Reduction
Keywords: Opioid Use Disorder; Harm Reduction; Peer Support; Peer Support Specialists
MeSH Terms: conditions — Opioid-Related Disorders; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Intervention (Experimental)
  Interventions: Behavioral: Peer Intervention
- Enhanced Usual Care (Other)
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Peer Intervention — Participants will receive one peer-led, in-person session boosted by weekly text messages over a 12-week period.
  Arms: Peer Intervention
Other: Enhanced Usual Care — Participants will receive a handout that includes harm reduction education and resources in their local area as part of enhanced usual care.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of the study is to develop an acceptable, feasible, and effective peer-led bundle of harm reduction services to be delivered in the hospital setting, called the THRIVE intervention.

The main question it aims to answer is: Will participants receiving the THRIVE intervention have a reduced risk of self-reported non-fatal overdoses OR skin/soft tissue infections compared to participants receiving enhanced usual care?

Researchers will compare the THRIVE model to enhanced usual care to see if the THRIVE model helps participants reduce their number of self-reported non-fatal overdoses OR skin/soft tissue infections.

Intervention participants will:

* Receive one in-person session from a peer support specialist while in the hospital
* Receive weekly text messages from the peer support specialist for a 12-week period
* Receive monthly, multiple-choice assessments via text message at Month 1, 2, 3, 4, 5, and 6
* Complete a baseline, 3-month, and 6-month assessment with Research Assistants

Enhanced usual care participants will:

* Receive a handout with harm reduction education and resources in their local area
* Receive monthly, multiple-choice assessments via text message at Month 1, 2, 3, 4, 5, and 6
* Complete a baseline, 3-month, and 6-month assessment with Research Assistants

ELIGIBILITY:
Inclusion Criteria:

* Participants who are: a) admitted to University of Pittsburgh Medical Center (UPMC) Shadyside Hospital, UPMC Presbyterian-Montefiore Hospital, UPMC Mercy Hospital for inpatient or observation status, or b) seen in the Emergency Department setting at UPMC Presbyterian-Montefiore Hospital and UPMC Mercy Hospital.
* Participants must have a current diagnosis of Opioid Use Disorder based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria.
* Participants must be at least 18 years of age on day of admission.
* Participants must be able to speak and read English.

Exclusion Criteria:

* Participants diagnosed with dementia and/or cognitive impairments.
* Participants with acute psychiatric complications, such as schizophrenia with acute psychosis, acute mania, or suicidal ideation (which may impact the ability of a participant to consent and actively participate in treatment).
* Participants who are pregnant or lactating at onset of study.
* Participants who cannot read or speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the THRIVE intervention compared to enhanced usual care (EUC) at lowering the incidence of non-fatal overdoses OR skin and soft tissue infections | Baseline to 6 months
  Cumulative incidence of non-fatal overdose OR skin and soft tissue infection

SECONDARY OUTCOMES:
Effectiveness of the THRIVE intervention compared to EUC at lowering the incidence of non-fatal overdoses | Baseline to 6 months
  Cumulative incidence of non-fatal overdose
Effectiveness of the THRIVE intervention compared to EUC at lowering the incidence of skin and soft tissue infections | Baseline to 6 months
  Cumulative incidence of skin and soft tissue infection

OTHER OUTCOMES:
Effectiveness of the THRIVE intervention on change in higher risk infection behaviors (characterized by BIRSI score) compared to EUC | Baseline to 6 months
  Change in higher risk infection behaviors measured as the total score on the BIRSI
Effectiveness of the THRIVE intervention on change in harm reduction adoption compared to EUC (a) | Baseline to 6 months
  (a) Change in the proportion of participants who self-report naloxone use in past 30 days to reverse another person's overdose
Effectiveness of the THRIVE intervention on change in harm reduction adoption compared to EUC (b) | Baseline to 6 months
  (b) Change in the proportion of participants who self-report currently carrying naloxone
Effectiveness of the THRIVE intervention on change in harm reduction adoption compared to EUC (c) | Baseline to 6 months
  (c) Change in the proportion of participants who self-report using at least one drug checking strategy in the past 30 days
Effectiveness of the THRIVE intervention on harm reduction access compared to EUC (a) | Baseline to 6 months
  (a) Change in the proportion of participants who self-report having received at least one of: naloxone, syringes, or new or unused pipes in past 30 days
Effectiveness of the THRIVE intervention on harm reduction access compared to EUC (b) | Baseline to 6 months
  (b) Change in the proportion of participants who self-report visiting a syringe services program in past 30 days
Effectiveness of the THRIVE intervention on harm reduction access compared to EUC (c) | Baseline to 6 months
  (c) Change in the proportion of participants who self-report receiving any harm reduction services from a needle exchange facility in past 30 days
Heterogeneity of treatment effect by race (Black versus white) in the THRIVE intervention arm | Baseline to 6 months
  Cumulative incidence of non-fatal overdose OR skin or soft tissue infection, by race (Black versus white)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline D Wilson, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian-Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harm Reduction Principles. National Harm Reduction Coalition. Accessed September 9, 2022. https://harmreduction.org/about-us/principles-of-harm-reduction/
- [Background] Friedman SR, de Jong W, Rossi D, Touze G, Rockwell R, Des Jarlais DC, Elovich R. Harm reduction theory: users' culture, micro-social indigenous harm reduction, and the self-organization and outside-organizing of users' groups. Int J Drug Policy. 2007 Mar;18(2):107-17. doi: 10.1016/j.drugpo.2006.11.006. Epub 2006 Dec 28. PMID 17689353
- [Background] Pauly BB, Reist D, Belle-Isle L, Schactman C. Housing and harm reduction: what is the role of harm reduction in addressing homelessness? Int J Drug Policy. 2013 Jul;24(4):284-90. doi: 10.1016/j.drugpo.2013.03.008. Epub 2013 Apr 25. PMID 23623720
- [Background] Pauly B, Wallace B, Barber K. Turning a blind eye: implementation of harm reduction in a transitional programme setting. Drugs Educ Prev Policy. 2018;25(1):21-30. doi:10.1080/09687637.2017.1337081
- [Background] Pauly B. Harm reduction through a social justice lens. Int J Drug Policy. 2008 Feb;19(1):4-10. doi: 10.1016/j.drugpo.2007.11.005. Epub 2008 Jan 15. PMID 18226520
- [Background] Stein MD, Phillips KT, Herman DS, Keosaian J, Stewart C, Anderson BJ, Weinstein Z, Liebschutz J. Skin-cleaning among hospitalized people who inject drugs: a randomized controlled trial. Addiction. 2021 May;116(5):1122-1130. doi: 10.1111/add.15236. Epub 2020 Sep 21. PMID 32830383
- [Background] Phillips KT, Stewart C, Anderson BJ, Liebschutz JM, Herman DS, Stein MD. A randomized controlled trial of a brief behavioral intervention to reduce skin and soft tissue infections among people who inject drugs. Drug Alcohol Depend. 2021 Apr 1;221:108646. doi: 10.1016/j.drugalcdep.2021.108646. Epub 2021 Feb 27. PMID 33677353
- [Background] Moustaqim-Barrette A, Dhillon D, Ng J, Sundvick K, Ali F, Elton-Marshall T, Leece P, Rittenbach K, Ferguson M, Buxton JA. Take-home naloxone programs for suspected opioid overdose in community settings: a scoping umbrella review. BMC Public Health. 2021 Mar 26;21(1):597. doi: 10.1186/s12889-021-10497-2. PMID 33771150
- [Background] McDonald R, Strang J. Are take-home naloxone programmes effective? Systematic review utilizing application of the Bradford Hill criteria. Addiction. 2016 Jul;111(7):1177-87. doi: 10.1111/add.13326. Epub 2016 Mar 30. PMID 27028542
- [Background] Krieger MS, Yedinak JL, Buxton JA, Lysyshyn M, Bernstein E, Rich JD, Green TC, Hadland SE, Marshall BDL. High willingness to use rapid fentanyl test strips among young adults who use drugs. Harm Reduct J. 2018 Feb 8;15(1):7. doi: 10.1186/s12954-018-0213-2. PMID 29422052
- [Background] Sherman SG, Morales KB, Park JN, McKenzie M, Marshall BDL, Green TC. Acceptability of implementing community-based drug checking services for people who use drugs in three United States cities: Baltimore, Boston and Providence. Int J Drug Policy. 2019 Jun;68:46-53. doi: 10.1016/j.drugpo.2019.03.003. Epub 2019 Apr 13. PMID 30991301
- [Background] Goldman JE, Waye KM, Periera KA, Krieger MS, Yedinak JL, Marshall BDL. Perspectives on rapid fentanyl test strips as a harm reduction practice among young adults who use drugs: a qualitative study. Harm Reduct J. 2019 Jan 8;16(1):3. doi: 10.1186/s12954-018-0276-0. PMID 30621699
- [Background] Peiper NC, Clarke SD, Vincent LB, Ciccarone D, Kral AH, Zibbell JE. Fentanyl test strips as an opioid overdose prevention strategy: Findings from a syringe services program in the Southeastern United States. Int J Drug Policy. 2019 Jan;63:122-128. doi: 10.1016/j.drugpo.2018.08.007. Epub 2018 Oct 3. PMID 30292493
- [Background] Hawk M, Coulter RWS, Egan JE, Fisk S, Reuel Friedman M, Tula M, Kinsky S. Harm reduction principles for healthcare settings. Harm Reduct J. 2017 Oct 24;14(1):70. doi: 10.1186/s12954-017-0196-4. PMID 29065896
- [Background] Chan CA, Canver B, McNeil R, Sue KL. Harm Reduction in Health Care Settings. Med Clin North Am. 2022 Jan;106(1):201-217. doi: 10.1016/j.mcna.2021.09.002. PMID 34823731
- [Background] Wilson JD, Berk J, Adger H, Feldman L. Identifying Missed Clinical Opportunities in Delivery of Overdose Prevention and Naloxone Prescription to Adolescents Using Opioids. J Adolesc Health. 2018 Aug;63(2):245-248. doi: 10.1016/j.jadohealth.2018.05.011. PMID 30149925
- [Background] Wilson JD, Spicyn N, Matson P, Alvanzo A, Feldman L. Internal medicine resident knowledge, attitudes, and barriers to naloxone prescription in hospital and clinic settings. Subst Abus. 2016 Jul-Sep;37(3):480-487. doi: 10.1080/08897077.2016.1142921. Epub 2016 Jan 28. PMID 26820604
- [Background] Deanna Wilson J, Berk J, Matson P, Spicyn N, Alvanzo A, Adger H, Feldman L. A Cross-sectional Survey Using Clinical Vignettes to Examine Overdose Risk Assessment and Willingness to Prescribe Naloxone. J Gen Intern Med. 2019 Apr;34(4):507-509. doi: 10.1007/s11606-018-4733-y. No abstract available. PMID 30406568
- [Background] Macalino GE, Sachdev DD, Rich JD, Becker C, Tan LJ, Beletsky L, Burris S. A national physician survey on prescribing syringes as an HIV prevention measure. Subst Abuse Treat Prev Policy. 2009 Jun 8;4:13. doi: 10.1186/1747-597X-4-13. PMID 19505336
- [Background] Stack E, Hildebran C, Leichtling G, Waddell EN, Leahy JM, Martin E, Korthuis PT. Peer Recovery Support Services Across the Continuum: In Community, Hospital, Corrections, and Treatment and Recovery Agency Settings - A Narrative Review. J Addict Med. 2022 Jan-Feb 01;16(1):93-100. doi: 10.1097/ADM.0000000000000810. PMID 33560695
- [Background] Mercer F, Miler JA, Pauly B, Carver H, Hnizdilova K, Foster R, Parkes T. Peer Support and Overdose Prevention Responses: A Systematic 'State-of-the-Art' Review. Int J Environ Res Public Health. 2021 Nov 17;18(22):12073. doi: 10.3390/ijerph182212073. PMID 34831839
- [Background] Kennedy MC, Boyd J, Mayer S, Collins A, Kerr T, McNeil R. Peer worker involvement in low-threshold supervised consumption facilities in the context of an overdose epidemic in Vancouver, Canada. Soc Sci Med. 2019 Mar;225:60-68. doi: 10.1016/j.socscimed.2019.02.014. Epub 2019 Feb 10. PMID 30798157
- [Background] Owczarzak J, Weicker N, Urquhart G, Morris M, Park JN, Sherman SG. "We know the streets:" race, place, and the politics of harm reduction. Health Place. 2020 Jul;64:102376. doi: 10.1016/j.healthplace.2020.102376. Epub 2020 Jul 22. PMID 32838893
- [Background] Bardwell G, Kerr T, Boyd J, McNeil R. Characterizing peer roles in an overdose crisis: Preferences for peer workers in overdose response programs in emergency shelters. Drug Alcohol Depend. 2018 Sep 1;190:6-8. doi: 10.1016/j.drugalcdep.2018.05.023. Epub 2018 Jun 26. PMID 29960202
- [Background] Pauly B, Wallace B, Pagan F, Phillips J, Wilson M, Hobbs H, Connolly J. Impact of overdose prevention sites during a public health emergency in Victoria, Canada. PLoS One. 2020 May 21;15(5):e0229208. doi: 10.1371/journal.pone.0229208. eCollection 2020. PMID 32438390
- [Background] Small W, Wood E, Tobin D, Rikley J, Lapushinsky D, Kerr T. The Injection Support Team: a peer-driven program to address unsafe injecting in a Canadian setting. Subst Use Misuse. 2012 Apr;47(5):491-501. doi: 10.3109/10826084.2012.644107. PMID 22428817
- [Background] Hayashi K, Wood E, Wiebe L, Qi J, Kerr T. An external evaluation of a peer-run outreach-based syringe exchange in Vancouver, Canada. Int J Drug Policy. 2010 Sep;21(5):418-21. doi: 10.1016/j.drugpo.2010.03.002. Epub 2010 Mar 31. PMID 20359877
- [Background] Dechman MK. Peer helpers' struggles to care for "others" who inject drugs. Int J Drug Policy. 2015 May;26(5):492-500. doi: 10.1016/j.drugpo.2014.12.010. Epub 2015 Jan 8. PMID 25630481
- [Background] Marshall C, Perreault M, Archambault L, Milton D. Experiences of peer-trainers in a take-home naloxone program: Results from a qualitative study. Int J Drug Policy. 2017 Mar;41:19-28. doi: 10.1016/j.drugpo.2016.11.015. Epub 2016 Dec 24. PMID 28027483
- [Background] Callon C, Charles G, Alexander R, Small W, Kerr T. 'On the same level': facilitators' experiences running a drug user-led safer injecting education campaign. Harm Reduct J. 2013 Mar 6;10:4. doi: 10.1186/1477-7517-10-4. PMID 23497293
- [Background] Colon RM, Deren S, Guarino H, Mino M, Kang SY. Challenges in recruiting and training drug treatment patients as peer outreach workers: a perspective from the field. Subst Use Misuse. 2010 Oct;45(12):1892-908. doi: 10.3109/10826081003684863. PMID 20380554
- [Background] Newland J, Treloar C. Peer education for people who inject drugs in New South Wales: Advantages, unanticipated benefits and challenges. Drugs Educ Prev Policy. 2013;20(4):304-311. doi:10.3109/09687637.2012.761951
- [Background] Hay B, Henderson C, Maltby J, Canales JJ. Influence of Peer-Based Needle Exchange Programs on Mental Health Status in People Who Inject Drugs: A Nationwide New Zealand Study. Front Psychiatry. 2017 Jan 18;7:211. doi: 10.3389/fpsyt.2016.00211. eCollection 2016. PMID 28149282
- [Background] Cacari-Stone L, Wallerstein N, Garcia AP, Minkler M. The promise of community-based participatory research for health equity: a conceptual model for bridging evidence with policy. Am J Public Health. 2014 Sep;104(9):1615-23. doi: 10.2105/AJPH.2014.301961. Epub 2014 Jul 17. PMID 25033119
- [Background] Adams SA, Heiney SP, Brandt HM, Wirth MD, Khan S, Johnson H, Davis L, Wineglass CM, Warren-Jones TY, Felder TM, Drayton RF, Davis B, Farr DE, Hebert JR. A comparison of a centralized versus de-centralized recruitment schema in two community-based participatory research studies for cancer prevention. J Community Health. 2015 Apr;40(2):251-9. doi: 10.1007/s10900-014-9924-9. PMID 25086566
- [Background] Burke JG, Jones J, Yonas M, Guizzetti L, Virata MC, Costlow M, Morton SC, Elizabeth M. PCOR, CER, and CBPR: alphabet soup or complementary fields of health research? Clin Transl Sci. 2013 Dec;6(6):493-6. doi: 10.1111/cts.12064. Epub 2013 May 8. PMID 24330697
- [Background] Horowitz CR, Brenner BL, Lachapelle S, Amara DA, Arniella G. Effective recruitment of minority populations through community-led strategies. Am J Prev Med. 2009 Dec;37(6 Suppl 1):S195-200. doi: 10.1016/j.amepre.2009.08.006. PMID 19896019
- [Background] Wilson JD, Altieri Dunn SC, Roy P, Joseph E, Klipp S, Liebschutz J. Inpatient Addiction Medicine Consultation Service Impact on Post-discharge Patient Mortality: a Propensity-Matched Analysis. J Gen Intern Med. 2022 Aug;37(10):2521-2525. doi: 10.1007/s11606-021-07362-8. Epub 2022 Jan 25. PMID 35076857
- [Background] Ojo SO, Bailey DP, Hewson DJ, Chater AM. Perceived Barriers and Facilitators to Breaking Up Sitting Time among Desk-Based Office Workers: A Qualitative Investigation Using the TDF and COM-B. Int J Environ Res Public Health. 2019 Aug 14;16(16):2903. doi: 10.3390/ijerph16162903. PMID 31416112
- [Background] McDonagh LK, Saunders JM, Cassell J, Curtis T, Bastaki H, Hartney T, Rait G. Application of the COM-B model to barriers and facilitators to chlamydia testing in general practice for young people and primary care practitioners: a systematic review. Implement Sci. 2018 Oct 22;13(1):130. doi: 10.1186/s13012-018-0821-y. PMID 30348165
- [Background] Timlin D, McCormack JM, Simpson EE. Using the COM-B model to identify barriers and facilitators towards adoption of a diet associated with cognitive function (MIND diet). Public Health Nutr. 2021 May;24(7):1657-1670. doi: 10.1017/S1368980020001445. Epub 2020 Aug 17. PMID 32799963
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Binswanger IA, Kral AH, Bluthenthal RN, Rybold DJ, Edlin BR. High prevalence of abscesses and cellulitis among community-recruited injection drug users in San Francisco. Clin Infect Dis. 2000 Mar;30(3):579-81. doi: 10.1086/313703. PMID 10722447
- [Background] Fink DS, Lindsay SP, Slymen DJ, Kral AH, Bluthenthal RN. Abscess and self-treatment among injection drug users at four California syringe exchanges and their surrounding communities. Subst Use Misuse. 2013 May;48(7):523-31. doi: 10.3109/10826084.2013.787094. Epub 2013 Apr 12. PMID 23581506
- [Background] Shrestha S, Stopka TJ, Hughto JMW, Case P, Palacios WR, Reilly B, Green TC. Prevalence and correlates of non-fatal overdose among people who use drugs: findings from rapid assessments in Massachusetts, 2017-2019. Harm Reduct J. 2021 Aug 30;18(1):93. doi: 10.1186/s12954-021-00538-9. PMID 34461922
- [Background] Stensrud MJ, Hernan MA. Why Test for Proportional Hazards? JAMA. 2020 Apr 14;323(14):1401-1402. doi: 10.1001/jama.2020.1267. No abstract available. PMID 32167523
- [Background] Bradburn MJ, Clark TG, Love SB, Altman DG. Survival analysis Part III: multivariate data analysis -- choosing a model and assessing its adequacy and fit. Br J Cancer. 2003 Aug 18;89(4):605-11. doi: 10.1038/sj.bjc.6601120. No abstract available. PMID 12915864